CLINICAL TRIAL: NCT02438033
Title: Characterizing the Specificity and Stability of Local Field Potentials in the Globus Pallidus Internus of Patients Undergoing Deep Brain Stimulation for Parkinson's Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Not approved by CMS
Sponsor: Nader Pouratian (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Nader Pouratian, Asst Professor of Neurosurgery, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PC PC+S
Record Dates: First submitted 2015-04-28; First posted 2015-05-08 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Parkinson's Disease
Keywords: Deep Brain Stimulation; Globus Pallidus; GPi; PC+S
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): All patients will be implanted with the investigational device in an open-label fashion
  Interventions: Device: Medtronic Activa PC+S Sensing Deep Brain Stimulator Generator

INTERVENTIONS:
Device: Medtronic Activa PC+S Sensing Deep Brain Stimulator Generator — Patients undergoing deep brain stimulation for Parkinson's disease based on clinically indicated criteria will have the option to enroll in this study, in which the Activa PC+S generator and corresponding extension leads will be implanted rather than the standard Activa PC system. Patients will be assessed every month for 3 months and then every 3 months after, including off and on medication assessments.

SUMMARY:
Deep brain stimulation for Parkinson's disease is a well established therapy. Current practice requires tedious adjustment of stimulation settings based on frequent patient assessments. Ultimately, the goal is to develop a system that can program itself using signals that are recorded directly from the brain on a continuous basis. Our previous work has identified abnormal electrical signals in the brain that are targeted for stimulation that can potentially be used to develop a self-programming system. In this study, the investigators will test the safety and utility of a novel adapted device that can not only deliver stimulation to the brain but also record brain signals in a patient that is implanted with a deep brain stimulation system. The purpose of this Phase I study is to understand the safety of the device as well as the relationship between these electrical signals measured from deep within the brain and Parkinson's symptoms and how these signals can be used to guide a self-programmed system. The study will entail implanting this special device (Activa PC+S) in place of the standard generator (Activa PC) and to compare clinical symptoms, recorded brain signals, and stimulation patterns during a one year period after implantation. Specifically, the investigators will use the Activa PC+S to record GPi (internal globus pallidus) local field potentials between and during programming visits, allowing the surgeon to better characterize a patient's disease. At the same time, the investigators will evaluate the safety of this new device.

DETAILED DESCRIPTION:
The device being tested is the Activa Primary Cell and Sensing (PC+S) system which consists of a deep brain stimulation (DBS) generator, specially adapted extension leads, and DBS leads implanted in the globus pallidus internus (GPi) in patients with Parkinson's disease (PD). The Activa PC+S system differs from currently FDA-approved devices in that it is not only capable of delivering therapeutic stimulation through the DBS leads but also recording electrophysiological signals through the same leads. The goal of this pilot study is to evaluate (1) to assess the specificity and stability of the electrophysiological signals recorded with the Activa PC+S system, (2) how the signals recorded by this system correlate with clinical parameters and non-invasive measures of movement, and (3) and the safety of the PC+S system.

The Medtronic Activa Primary Cell (PC) DBS system has a proven record of safety and reliability through extensive human clinical use over the years1. The potential risks associated with the placement and the use of the device have been thoroughly described in previous human trials and retrospective reports. The PC+S device is based on the currently approved device but with added sensing capabilities. In this protocol, we will evaluate the Activa PC+S system using additional sensing components with stimulation parameters commonly used for the treatment of movement disorder.

This trial will follow a non-randomized design with rigorous and comprehensive follow-ups, as described below.

The study will be conducted at the Ronald Reagan UCLA Medical Center and associated facilities through the combined neurology and neurosurgery movement disorders program, which manages over 1,000 patients with PD. The study will provide close follow-up of patients after DBS surgery by a team involving functional neurosurgeons and neurologists with expertise in clinical care of patients with PD.

Patients will be screened according to the inclusion/exclusion criteria. Each patient will be informed about the study to see if they are interested in participating. After the patient signs the informed consent, they will undergo baseline evaluations, and if they qualify, they will undergo surgery to implant the deep brain stimulation system.

After device implantation, patients will complete comprehensive follow-up as described in the protocol below. The patients will return to the clinic at least monthly for the first 3 months for on and off medication assessments and programming. Primary assessments will be administered monthly for the first 3 months, and then every 3 months up to 12 months post-operatively.

LFPs will be recorded across time (intraoperative, during programming, and chronically), across activity states (with quantitative accelerometer and gyroscope measurements), and across disease states (off and on medication, off and on stimulation) to address the primary research questions proposed.

A comparison of measures within the same person from pre-treatment to post-treatment will be performed. Also, pre-treatment and post-treatment group means and standard deviations will be determined. Correlations between LFP biosignals and non-invasive measures and clinical assessment of movement will be performed. In addition, correlation between LFP signals and clinically-defined stimulation parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Chart diagnosis of PD as the principal neurologic diagnosis with evidence of dopamine responsiveness.
2. Documented PD duration > 5 years.
3. Clinical indications for GPi DBS based on presence of motor fluctuations with troublesome dyskinesias despite best medical therapy.
4. Age ≥ 21 years of age.
5. Able to give informed consent in accordance with institutional policies and participate in the 1-year follow-up, involving assessments and stimulator adjustments.
6. Willingness to have unexpected neurological or psychiatric symptoms shared with study clinicians.
7. Other medical conditions must be stable for at least 1 year, (conditions that require intermittent use of steroids or chemotherapy are excluded).

Exclusion Criteria:

1. Tremor-dominant PD.
2. Significant neurocognitive impairment in memory domain suggestive of dementing process (based on MOCA and PD-CRS, described below).
3. Age > 75 years.
4. History of implant-related infection.
5. History of bleeding or immune-compromise.
6. Patient living greater than 100 miles from UCLA.
7. Suicide attempt in the last two years and/or presence of a suicide plan (an answer of "Yes" to Question C4 in Section C-Suicidality of MINI International Neuropsychiatric Interview).
8. Alcohol or illicit substance use disorder within the last 6 months, unstable remission of substance abuse, or chart evidence that co-morbid substance use disorder could account for lack of treatment response.
9. Current significant neurological conditions, including epilepsy, stroke, or history of serious head injury with loss of consciousness.
10. Uncontrolled medical condition including cardiovascular problems and diabetes.
11. Pregnant or planning to become pregnant
12. Uncontrolled chronic pain.
13. Preoperative use of warfarin or any blood thinning or antiplatelet agent or any patient with abnormally elevated preoperative coagulation profile (either PTT or PT/INR)..
14. Significant abnormality on preoperative structural brain MRI.
15. Contraindications to MRIs or the need for recurrent body MRIs.
16. High risk for surgery.
17. Has cardiac pacemaker/defibrillator, implanted medication pump, intra-cardiac lines, any intracranial implants (e.g., aneurysm clip, shunt, cochlear implant, electrodes) or other implanted stimulator.
18. Patient has had past cranial neurosurgery.
19. Patient unable to discontinue therapeutic diathermy.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Change in Unified Parkinson's Disease Rating Scale (UPDRS) | 12 months

SECONDARY OUTCOMES:
Change in Hoehn and Yahr Scale | 12 months
Change in Parkinson's Disease Questionnaire (PDQ-39) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nader Pouratian, MD PhD, Principal Investigator — University of California, Los Angeles